CLINICAL TRIAL: NCT07142031
Title: In-Vivo Application and Clinical Evaluation of Onlay Restorations Fabricated From BioHPP Polymer and Lithium Disilicate Ceramic Materials
Brief Title: BioHPP and Lithium Disilicate Onlay Restorations: Clinical Evaluation
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Ege University (Other)
Collaborators: The Scientific and Technological Research Council of Turkey (Other)
Responsible Party: Principal Investigator, Ayşe Gözde Türk, Associate Prof., Ege University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Other
Other Study IDs: Ege-DHF-AGT-01
Record Dates: First submitted 2025-08-19; First posted 2025-08-26 (Actual); Last update posted 2025-11-14 (Actual); Status verified 2025-11

CONDITIONS: Dental Caries; Polymers
Keywords: Polyetheretherketones; Dental Porcelain; Dental Restoration, permanent; Computer-Aided Design
MeSH Terms: conditions — Dental Caries | interventions — lithia disilicate

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Masking Description: To eliminate predictability and minimize any potential bias, the first group will be determined using the coin toss randomization method, followed by the application of block randomization in blocks of four. After the initial four patients in the first group are completed, patient allocation to the second group will proceed in blocks of four, and the distribution of all participants will be completed according to block randomization. Neither the patients included in the study nor the evaluator will be aware of the group assignments, with only the principal investigator having knowledge of the allocation.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- BioHPP Onlay Restorations: Clinical Evaluation (Experimental): The onlay preparation for the designated tooth of each patient included in the study will be performed using an onlay preparation bur set under water cooling with a rotary handpiece. Subsequently, digital impressions of the prepared teeth will be obtained using an intraoral scanner to facilitate the design of the onlay restorations. Following their design and fabrication, the BioHPP onlay restorations will be adhesively cemented to the teeth after verifying their fit.
  Interventions: Other: BioHPP
- Lithium Disilicate Onlay Restorations: Clinical Evaluation (Active Comparator): The onlay preparation for the designated tooth of each patient included in the study will be performed using an onlay preparation bur set under water cooling with a rotary handpiece. Subsequently, digital impressions of the prepared teeth will be obtained using an intraoral scanner to facilitate the design of the onlay restorations. Following their design and fabrication, the Lithium Disilicate onlay restorations will be adhesively cemented to the teeth after verifying their fit.
  Interventions: Other: Lithium Disilicate

INTERVENTIONS:
Other: BioHPP — Onlay restorations fabricated from BioHPP polymer will be applied to 20 patients. Following the 6- and 12-month follow-ups, the collected data will be analyzed according to clinical evaluation criteria.
  Arms: BioHPP Onlay Restorations: Clinical Evaluation
Other: Lithium Disilicate — Onlay restorations fabricated from lithium disilicate will be applied to 20 patients and will serve as the control group for comparison with the BioHPP onlay restorations. Following the 6- and 12-month follow-ups, the collected data will be analyzed according to clinical evaluation criteria.
  Arms: Lithium Disilicate Onlay Restorations: Clinical Evaluation

SUMMARY:
In this study, clinical data obtained from the in vivo evaluation of onlay restorations fabricated with CAD/CAM using modified PEEK (BioHPP Shade 2, Bredent group GmbH & Co. KG, Senden, Germany) and lithium disilicate (IPS e.max CAD, Ivoclar Vivadent, Schaan, Liechtenstein) ceramic materials will be analyzed, and the clinical outcomes will be assessed to investigate the clinical applicability of BioHPP. The clinical success of the restorations will be evaluated using established clinical evaluation criteria, specifically the modified United States Public Health Service (USPHS) criteria, focusing on parameters such as marginal adaptation, surface roughness, color match, anatomical form, and participant-reported outcomes. These restorations will be applied to molar teeth in the maxilla and mandible, provided that the teeth are vital and have no adjacent or opposing restorations. Only teeth meeting these inclusion criteria will be considered in the study.

DETAILED DESCRIPTION:
Patients aged between 18 and 50 years, systemically healthy, with good oral hygiene, without periodontal disease, and with at least 24 teeth present in the oral cavity (including the first permanent molars) to ensure balanced occlusal load distribution during mastication, will be included. Only patients without parafunctional habits or smoking, and in whom esthetic criteria are not a primary concern, will be enrolled. The treated tooth must be vital, with intact buccal and lingual enamel walls measuring 2-3 mm in thickness, while the mesial and distal surfaces are destroyed. Additionally, the presence of a MOD (mesio-occluso-distal) preparation in which the isthmus involves more than half of the buccolingual width of the tooth, and the tooth does not require full crown restoration, will be required. Eligible teeth include the maxillary right and left first molars (teeth 16 and 26) and second molars (teeth 17 and 27), as well as the mandibular right and left first molars (teeth 46 and 36) and second molars (teeth 47 and 37).

For standardization purposes, the onlay cavity preparation will be restricted to cases in which the buccal and lingual enamel walls remain 2-3 mm in thickness, and the isthmus covers more than half of the buccolingual width of the tooth. If these limits are exceeded during cavity preparation or if pulp perforation occurs, the necessary treatment will be provided for the respective tooth, but such cases will be excluded from the study.

The aim of the study is to overcome the limitations of in vitro studies, such as the inability to replicate intraoral conditions (oral aging, fatigue stress, diet, and microtrauma), by evaluating BioHPP onlay and lithium disilicate restorations in vivo with respect to parameters including color match, marginal discoloration, anatomical form, marginal adaptation, surface texture, and fracture. The purpose of the project is to investigate the clinical success of onlay restorations fabricated using Computer-Aided Design/Computer-Aided Manufacturing (CAD/CAM) with BioHPP and lithium disilicate ceramic (IPS e.max CAD) materials.

ELIGIBILITY:
Inclusion Criteria:

* The teeth planned for onlay restoration (teeth numbered 16, 17, 26, 27, 36, 37, 46, and 47) with destroyed mesial and distal surfaces, but with intact buccal and lingual enamel walls of 2-3 mm thickness.
* In the tooth to be treated, the presence of a MOD (mesio-occluso-distal) preparation where the isthmus involves more than half of the buccolingual width of the tooth, or where the distance between the fissure and cusp tip exceeds one-third of the intercuspal distance, including one or more cusps.
* Teeth that do not require full crown restoration.
* Absence of any other restorations on the adjacent teeth (mesial/distal) or on the opposing teeth corresponding to the tooth planned for onlay restoration.
* Since the BioHPP polymer material used in this study is not an esthetic material and does not offer color options, only posterior teeth that do not pose esthetic concerns will be included: maxillary right and left first molars (teeth 16 and 26) and second molars (teeth 17 and 27), as well as mandibular right and left first molars (teeth 46 and 36) and second molars (teeth 47 and 37).

Exclusion Criteria:

* The relevant tooth being non-vital
* Presence of crowns on the adjacent (mesial and distal) or opposing teeth
* Absence of proper occlusal contact of the relevant tooth
* Patient having periodontitis
* Patient age not within the 18-50 year range
* Presence of bruxism in the patient

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 40 (Estimated)
Dates: Start 2025-09-15 (Actual); Primary Completion 2026-09-15 (Estimated); Study Completion 2026-10-15 (Estimated)

PRIMARY OUTCOMES:
Modified United States Public Health Service (USPHS) Criteria | one year
  The clinical performance of the onlay restorations was evaluated using the modified USPHS (United States Public Health Service) criteria. Parameters such as color match, anatomic form, marginal integrity, surface roughness, retention, and postoperative sensitivity were assessed. Each parameter was scored using Alpha, Bravo, and Charlie ratings, where Alpha indicates optimal clinical performance, Bravo represents an acceptable level, and Charlie denotes the need for restoration correction or replacement. In this system, higher scores correspond to better clinical performance, while lower scores indicate decreased performance.

CONTACTS AND LOCATIONS:
Locations (1):
- Ege University Faculty of Dentistry, Izmir, Bornova, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No
The sharing of patient data was not deemed necessary.